CLINICAL TRIAL: NCT06117761
Title: Combined Activity and Cognitive Intervention to Optimize Recovery From Critical Illness in ICU Survivors: COMBAT-ICU Trial
Brief Title: Combined Activity and Cognitive Intervention for ICU Survivors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW23-271
Record Dates: First submitted 2023-10-15; First posted 2023-11-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Post Intensive Care Syndrome; ARDS: Acute Respiratory Distress Syndrome; Delirium; Loss of Muscle Mass; Loss of Muscle Strength; Cognitive Function
Keywords: Post-intensive care syndrome; PICS; Intensive Care Unit; ICU survivors; home-based exercise
MeSH Terms: conditions — postintensive care syndrome; Acute Lung Injury; Delirium | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COMBAT-ICU (Experimental): The COMBAT-ICU group will receive an intervention which will last for 8 weeks, with 3 sessions per week. A blended training platform with supervised in-person home visits and a real-time supervised online and unsupervised selfpractice approach will be used to deliver the intervention, with the platform gradually shifted from home visits to unsupervised self-practice according to participants' physical functioning level. Family caregivers will be involved in the intervention, so that they can facilitate home-based training. Each intervention session will last for 80 minutes and comprise 45 minutes of exercise training, a 5-minute break and 30 minutes of cognitive training. Moreover, all participants in the COMBAT-ICU group will be invited to complete a satisfaction survey and semi-structured qualitative interview, which will focus on exploring the acceptability and perceived effects from participants' perspective.
  Interventions: Other: Home-based exercises combined with cognitive training
- Exercise Group (Experimental): The exercise group will receive an 8-week, home-based, exercise intervention which is the same as that of the exercise component of the COMBAT-ICU intervention, 3 sessions per week, and 45 minutes per session, but will not receive any structured cognitive training.
  Interventions: Other: Home-based exercises
- Attention Placebo Group (Placebo Comparator): The attention placebo group will receive a telephone call every 2 weeks, with the conversation focused on information provision and brief counselling relating to their health conditions, in order to reduce the potential bias from greater attention for the COMBAT-ICU and exercise groups. They will also receive the routine care provided by the healthcare system, including medical follow-ups with the clinical team, without structured out-patient rehabilitation services.
  Interventions: Other: Attention Placebo

INTERVENTIONS:
Other: Attention Placebo — Telephone follow-up focused on information provision and brief counselling relating to their health conditions. They will also receive routine care from the healthcae system, including medical follow-ups with the clinical team, without structured out-patient rehabilitation services.
  Arms: Attention Placebo Group
Other: Home-based exercises combined with cognitive training — An 8-week, home-based, exercise with cognitive training intervention. 3 sessions per week, and 80 minutes per session.It comprises of 45 minutes of exercise training, a 5-minute break and 30 minutes of cognitive training.A blended training platform with supervised in-person home visits and a real-time supervised online and unsupervised selfpractice approach will be used to deliver the intervention, with the platform gradually shifted from home visits to unsupervised self-practice according to participants' physical functioning level. Family caregivers will be involved in the intervention, so that they can facilitate home-based training. Each intervention session will last for 80 minutes and comprise 45 minutes of exercise training, a 5-minute break and 30 minutes of cognitive training.
  Arms: COMBAT-ICU
Other: Home-based exercises — An 8-week, home-based, exercise-only intervention. Weeks 1 and 2 will be the induction phase, all sessions will be supervised with two home visit sessions and one online session in real-time. Weeks 3 to 6 will be the maintenance phase. For participants with a higher functional performance level (Level 3 or 4), the mode of delivery will change to one home visit and two online training sessions. Weeks 7 and 8 will be the consolidation phase, consisting of two online sessions and one unsupervised self-practice session. They will not receive any structured cognitive training.
  Arms: Exercise Group

SUMMARY:
This mixed-methods study comprising a 3-arm pilot RCT and a qualitative study aims to investigate the preliminary effects and feasibility of a home-based combined activity and cognitive intervention for ICU survivors (COMBAT-ICU). Adopting a 3-arm design with COMBAT-ICU, exercise and attention placebo study arms will enable us to evaluate the added effects, if any, of the novel combined intervention compared with the standard exercise-only rehabilitation strategy and attention placebo. Data triangulation from quantitative and qualitative aspects can facilitate result interpretation. The study's objectives are:

1. To evaluate the preliminary effects of the COMBAT-ICU intervention for ICU survivors on PICS, physical, mental and cognitive outcomes, HRQoL, unplanned re-hospitalisation rate, and mortality.
2. To explore the feasibility and acceptability of the COMBAT-ICU intervention and ICU survivors' intervention engagement experience.

The hypothesis of the first objective is that upon completion of the COMBAT-ICU intervention, ICU survivors will have reduced PICS, improved physical function, mental health, cognition and HRQoL, and reduced unplanned readmissions and mortality compared with the exercise and attention placebo groups at post-intervention and 3 months thereafter. While the hypothesis of the second objective is that the COMBAT-ICU intervention is feasible and acceptable for ICU survivors.

DETAILED DESCRIPTION:
With the growing cohort of patients surviving after ICU treatment, the long-term consequences of critical illness have gained increased attention in the past decade. It is common for ICU survivors to experience long-term impairments in one or more domains of physical, cognitive or psychological functioning that persist beyond acute care hospitalization for a critical illness, impairments that are collectively known as post-intensive care syndrome (PICS).

As PICS is a relatively new syndrome, research is accumulating on different approaches to tackling it. There are several limitations on previous studies, such as only a single strategy, an exercise intervention, was tested to manage physical impairment or PICS as a whole, or no beneficial effect was documented on health-related QoL, leaving a significant gap in the literature. Hence, a multimodal rehabilitative approach is needed for this vulnerable cohort in promoting physical, functional and cognitive performance so as to develop effective strategies to prevent and manage PICS among ICU survivors, particularly during the early post-discharge period.

This study is mixed-methods comprising a 3-arm pilot RCT and a qualitative study aims to investigate the preliminary effects and feasibility of a home-based combined activity and cognitive intervention for ICU survivors (COMBAT-ICU), with assessments measured at baseline, immediate post-intervention and 3 months post-intervention. It will be conducted in three public hospitals in Hong Kong. Patients fulfilling the following eligibility criteria will be recruited: 1) Chinese adults aged ≥18; 2) has been admitted to ICU for at least 4 days; 3) has been discharged home; 4) was able to perform basic activities of daily living before ICU admission; 5) is living with family; 6) has an electronic device that can access the internet (patient/family); 7) is able to walk for at least 10 metres (assisted or unassisted).

Participants will be randomly allocated in a 1:1:1 ratio to the COMBAT-ICU, exercise or attention placebo groups.

For the COMBAT-ICU group, they will receive an intervention which will last for 8 weeks, with 3 sessions per week. A blended training platform with supervised in-person home visits and a real-time supervised online and unsupervised self practice approach will be used to deliver the intervention, with the platform gradually shifted from home visits to unsupervised self-practice according to participants' physical functioning level. Family caregivers will be involved in the intervention, so that they can facilitate home-based training. Each intervention session will last for 80 minutes and comprise 45 minutes of exercise training, a 5-minute break and 30 minutes of cognitive training. Moreover, all participants in the COMBAT-ICU group will be invited to complete a satisfaction survey and semi-structured qualitative interview, which will focus on exploring the acceptability and perceived effects from participants' perspective.

For the exercise group, they will receive an 8-week, home-based, exercise intervention which is the same as that of the exercise component of the COMBAT-ICU intervention, 3 sessions per week, and 45 minutes per session, but will not receive any structured cognitive training.

For the attention placebo group, they will receive a telephone call every 2 weeks, with the conversation focused on information provision and brief counselling relating to their health conditions, in order to reduce the potential bias from greater attention for the COMBAT-ICU and exercise groups. They will also receive the routine care provided by the healthcare system, including medical follow-ups with the clinical team, without structured out-patient rehabilitation services.

Evaluative outcomes will be measured at baseline (T0), immediate post-intervention (T1) and 3 months post-intervention (T2), and include Post-Intensive Care Syndrome Questionnaire (PICSQ), muscle mass and strength, physical performance, cognition function, psychological distress, Health-related quality of life (HRQoL), hospital readmission and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged ≥18
2. has been admitted to ICU for at least 4 days
3. discharged home
4. able to perform basic activities of daily living before ICU admission
5. living with family
6. has an electronic device that can access the internet (patient/family)
7. able to walk for at least 10 metres (assisted or unassisted)

Exclusion Criteria:

1. cannot read Chinese
2. has musculoskeletal injury precluding exercise training
3. is receiving structured out-patient pulmonary or cardiac rehabilitation after discharge
4. has clinically evident dementia or significant impairment from an acute brain problem (e.g. traumatic brain injury, stroke, subarachnoid haemorrhage or hypoxic brain injury) that precludes following the study protocol
5. has prolonged length of stay (≥28 days) in the step-down wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported PICS | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The 18-item Post-Intensive Care Syndrome Questionnaire (PICSQ) will be used to measure the extent of PICS. The PICSQ consists of 3 subscales, physical, cognitive and mental, and is rated on a 4-point Likert scale ranging from 0 to 3. It has good internal consistency (Cronbach's alpha = 0.93). Its criterion validity is evidenced by its strong correlation with frailty and HRQoL measures, and factor analysis confirmed its construct validity.

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  6MWT will be used to evaluate aerobic capacity and endurance. Standard measurement guidelines will be followed, and the distance walked will be recorded.
Time-Up-Go test | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  Time-Up-Go test will be used to measure functional mobility, assessed by the time it takes to stand up, walk a distance of 10 feet, turn, walk back and sit down.
Short Physical Performance Battery | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The Short Physical Performance Battery will be used to assess functional capacity. It consists of 3 timed tasks: standing balance, walking speed and chair stand tests.
Grip strength | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  Handgrip strength will be assessed by a dynamometer to evaluate muscle strength of upper limbs.
Digit Span test | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The Digit Span test will be used to measure short-term and working memory.
Colour Trails Test | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  Colour Trails Test to measure executive function and attention. It has two parts: part 1 assesses visual-motor processing speed and attention, and part 2 sequencing and mental flexibility in addition to processing speed and attention.
Montreal Cognitive Assessment | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The Montreal Cognitive Assessment will be used to assess global cognition
Patient Health Questionnaire-9 | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The Patient Health Questionnaire-9 will be used to measure the frequency of depressive symptoms in the past 14 days. Its 9 items are rated on a 4-point scale ranging from 0 to 3, with higher sum scores indicating more depressive symptoms.
Generalized Anxiety Disorder Scale-7 | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  The Generalized Anxiety Disorder Scale-7 will be used to measure anxiety levels. Ratings on a 4-point scale (0-3) indicate the frequency of anxiety symptoms in the past 14 days, with higher total scores representing greater anxiety.
  HRQoL: The EuroQol Five Dimensions Five Levels (EQ-5D-5L) will be used to measure HRQoL. It consists of two parts: EQ-5D descriptive system and EQ visual analogue scale. The first part uses 5 levels to indicate a participant's health state on 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression - and the second part is an additional self-rated health item rated on a visual analogue scale ranging from 0-100.
EuroQol Five Dimensions Five Levels (EQ-5D-5L) | At baseline (T0), immediate post-intervention: 8 weeks (T1) and 3 months post-intervention (T2)
  EQ-5D-5L will be used to measure health-related quality of life. It consists of two parts: EQ-5D descriptive system and EQ visual analogue scale. The first part uses 5 levels to indicate a participant's health state on 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression - and the second part is an additional self-rated health item rated on a visual analogue scale ranging from 0-100.
Unplanned hospital readmission | From baseline (T0) to 3 months post-intervention (T2)
  Hospital utilisation data will be monitored from T0 to T2 through electronic medical record review.
mortality | From baseline (T0) to 3 months post-intervention (T2)
  mortality will be monitored from T0 to T2 through electronic medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Dr, Principal Investigator — The University of Hong Kong, School of Nursing
Locations (1):
- The School of Nursing, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT06117761/Prot_000.pdf